CLINICAL TRIAL: NCT01327768
Title: Evaluation of Safety, Feasibility and Treatment Potential for Old Stroke Patients Using Intracerebral Implantation of Olfactory Ensheathing Cells
Brief Title: Implantation of Olfactory Ensheathing Cells (OECs)
Acronym: OECs
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CN1U00-1
Record Dates: First submitted 2011-01-31; First posted 2011-04-04 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Infarction, Middle Cerebral Artery; Ischemic Stroke,; Stroke With Hemiparesis,; Thromboembolic Stroke.
Keywords: Stroke,; Stem Cell,; Olfactory Ensheathing Cells,; Intracerebral Implantation of Olfactory Ensheathing Cells.
MeSH Terms: conditions — Infarction, Middle Cerebral Artery; Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OECs, Medicine, Rehabilitation (Experimental): Stroke patients are received intracerebral implantation of Olfactory ensheathing cells(OECs), Antiplatelet Medication, and Rehabilitation.
  Interventions: Procedure: Olfactory ensheathing cells

INTERVENTIONS:
Procedure: Olfactory ensheathing cells — Recruited patients should be received the endoscopic surgery for picking the olfactory mucosa 1 to 2 months before transplantation. The OECs will be cultured and expanded under the rule of GTP. Finally, we will transplant the OECs (about 2 to 8 X 10´6 cells in saline) into the peri-infarcted area of the brain for old stroke ischemic patients.
  Other Names: Stroke,; Stem Cells,; Olfactory Ensheathing Cells,; Early Phase Clinical Trial.

SUMMARY:
Recruited patients should receive the endoscopic surgery for picking the olfactory mucosa 1 to 2 months before transplantation. The Olfactory Ensheathing Cells (OECs) will be cultured and expanded under the rule of GTP. Then, quality control of OECs should be done by immunohistochemical staining positive for GFAP, S100, and P75. Finally, the investigators will transplant the OECs (about 2 to 8 X 10´6 cells in saline) into the peri-infarcted area of the brain.

DETAILED DESCRIPTION:
(1)Recruited patients should receive the endoscopic surgery for picking the olfactory mucosa 1 to 2 months before transplantation. The OECs will be cultured and expanded under the rule of GTP. Then, quality control of OECs should be done by immunohistochemical staining positive for GFAP, S100, and P75. Finally, the investigators will transplanted the OECs (about 2 to 8 X 10´6 cells in saline) into the peri-infarcted area of the brain. (2) Combination with traditional drug therapy (such as used the anti-thrombosis reagent or anti-platelet aggregation reagent). (3) NIH-stroke scale (NIHSS), European stroke scale (ESS), European stroke motor subscale (EMS), Barthel Index(BI) and MMSE will be performed for each patient to evaluate the therapeutic effect as the primary end points. (4) In addition, MRI(DTI) & TMS(MEP) will be also checked for each recruitment patient as the secondary end points.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35-70 year old Chronic Stroke Adult Patients,
* With Stroke History of More Than 6 Months, Less Than 60 Months,
* With Stable Hemiplegia Condition,
* NIHSS Score Is Between 5~15.

Exclusion Criteria:

* Patients Aged Less Than 35 or More Than 70,
* Hemorrhage Stroke or MRI Show The Occlusion Is Not In The Middle Cerebral Artery Territory,
* NIHSS Is Not In The Range of 5~15,
* Pregnant Women,
* Impaired Liver Function, Abnormal Blood Coagulation, AIDS Carrier, Tumors, Other Special Conditions, etc.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
NIH-Stroke Scale | within 1 year after surgery
  National Institute of Health-Stroke Scale will be performed to evaluate including muscle power of hemiparetic limbs, sensory function and flurency of speech of each patient to document the therapeutic effect.

SECONDARY OUTCOMES:
MRI(DTI) | within 1 year after surgery
  Magnetic Resonance Image (Diffusion Tensor Image) will be performed to evaluate the increase of the number of fiber tracts (pyramidal tract) in the stroke brain of each patient to document the therapeutic effect.
TMS(MEP) | within 1 year after surgery
  Trans-cranial Magnetic Stimulation (Motor Evoked Potential) will be performed to evaluate the electrophysiological response of stroke brain of each patient to document the therapeutic effect.

CONTACTS AND LOCATIONS:
Overall Officials: Woei-Cherng Shyu, M.D., Ph.D, Study Chair — shyu9423@gmail.com
Locations (1):
- China Medical University Hospital, Center of Neuropsychiatry, Taichung, Taiwan